CLINICAL TRIAL: NCT05077514
Title: Increasing Treatment Seeking Among At-Risk Service Members Returning From Warzones
Brief Title: Treatment Seeking Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tracy Stecker, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00053847; W81XWH-13-2-032 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Behavioral: Experimental: Cognitive Behavior Therapy
- Group B (Active Comparator)
  Interventions: Behavioral: Active comparator: National Crisis Line

INTERVENTIONS:
Behavioral: Experimental: Cognitive Behavior Therapy — Participants assigned to Group A were asked to participate in a talking session with a psychologist regarding thoughts about treatment. This session is designed to explore thoughts about behavioral health therapy for suicidality. The session was administered by phone, initially and again one month later. Participants discussed current functioning and their thoughts about seeking help with the goal of modifying thoughts about treatment. This phone session lasted approximately 45 to 60 minutes.
  Arms: Group A
Behavioral: Active comparator: National Crisis Line — Participants assigned to Group B received information about the VA's National Crisis Line.
  Arms: Group B

SUMMARY:
The study team conducted a randomized controlled clinical trial of 809 military service members who were at increased risk for suicide but not currently in behavioral health treatment. This study tested the effectiveness of a brief phone-based intervention (CBT-TS) aimed at changing military member's perceptions about behavioral health therapy. Participants completed five interviews over the course of one year to collect information about change in behavioral health symptoms and treatment utilization.

DETAILED DESCRIPTION:
Participants A randomized controlled trial design was used to test the efficacy of a brief, manualized, evidence-based CBT-TS to promote treatment initiation among at-risk military members and Veterans (W81XWH-13-2-0032; Increasing Treatment Seeking among At-Risk Service Members Returning from Warzones, funded by the Department of Defense). Participants were recruited through media advertisements. Ads targeted individuals who were considering help seeking. Eligible participants: 1) served in the US Armed Forces after September 11, 2001, 2) were not receiving behavioral health treatment at the time of the screening, and 3) endorsed recent suicidal ideation on the PHQ-9, item 9 (i.e., score of 1 or higher on the item) or a lifetime suicide attempt. Study procedures were reviewed and approved by the appropriate institutional review boards.

Procedures Individuals deemed eligible after screening and who agreed to participate went through the informed consent process and were randomly assigned to either the control or CBT-TS condition. Participants were administered the baseline assessment with follow-up symptom and treatment utilization assessments occurring at months 1, 3, 6, and 12. All assessments were administered by telephone. Participants were compensated $25 for each assessment.

Conditions:

Cognitive Behavioral Treatment for Treatment Seeking. CBT-TS is a brief, manualized, phone-delivered, individual session lasting 45-60 minutes. CBT-TS targets a change in beliefs that influence whether someone enters treatment. A CBT-TS session has 4 distinct, successive stages. First, participants identify current symptoms. Second, participants describe strategies to manage symptoms. Third, beliefs about treatment are elicited. Fourth, participants discuss each stated belief. All participants were administered the same structured intervention; however, content discussed was personalized. For example, while participants may endorse similar beliefs about getting help (e.g., "Going to treatment would mean I am weak"), their ideas surrounding that belief and the meaning of it may differ. Therefore, while the intervention was structured, it allows for a personalized, tailored approach.

Control condition. Participants assigned to the control condition did not receive the CBT-TS session. They were administered assessment measures at all time points comparable to the experimental group.

Measures Demographic variables were assessed at baseline using a structured questionnaire.

The Perceptions about Services Scale (PASS) was administered at baseline and is a 28-item self-report measure assessing beliefs about treatment and the extent to which they intend to initiate treatment. The PASS was originally developed to inform the development of the CBT-TS intervention and has good test-retest reliability.

Measures of suicidal ideation, history of suicide attempt, and a range of clinical risk factors for suicidal ideation and behavior were obtained at baseline assessment to describe the sample, to facilitate a comparison of the CBT-TS and control group, and to guide any statistical adjustments that may be needed in the event of differences between groups. Suicidal ideation and suicide attempt were measured with the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS is a widely used and validated semi-structured, rater-based interview designed to assess the severity and frequency of current and past suicidal ideation and behaviors. The C-SSRS has strong psychometric properties, has been validated for administration by phone, and has been used in prior research of suicidal behavior in Veterans. Clinical risk factors for suicidal thoughts and behavior were assessed using validated, widely used, brief, structured questionnaires including assessments of: the number of days of alcohol use (5+ drinks) and non-prescribed drug use in the past 30 days (Addiction Severity Index - Alcohol and Drug Scales [ASI];, pain, sleep disturbance (Insomnia Severity Index), thwarted belonging and perceived burdensomeness (Interpersonal Needs Questionnaire), depressive symptoms (Patient Health Questionnaire-9) and post-traumatic stress disorder symptoms (PTSD Checklist for DSM-IV Military Version2).

Treatment utilization was assessed at months 1, 3, 6 and 12. There were two primary outcomes, treatment initiation to address suicidality or related conditions and the number of treatment sessions attended. Treatment initiation was assessed by asking participants if they had attended a mental health appointment. Data were collected as to the nature of the appointment, reason for the visit, whether they reported seeing a physician, psychologist, or other professional, and whether the session occurred at a VA facility or outside of VA. The other primary outcome, treatment sessions attended, was assessed by asking participants how many mental health treatment sessions they had attended.

Logistic regression was used to assess treatment initiation, a categorical outcome. Latent growth curve modeling was conducted to assess treatment sessions attended, a continuous outcome.

ELIGIBILITY:
Inclusion Criteria:

* Must be in US Military current or previous after September 11, 2001
* Must indicate suicidal ideation with in the past 2 weeks or have previous suicide attempt
* Not currently receiving behavioral health treatment

Exclusion Criteria:

* No suicide ideation or history of attempt
* currently receiving behavioral health treatment

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 809 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Change in attitudes towards behavioral health treatment | 1 month after intervention
  Change in mean score on the Perceptions about Services Scale (a measure of attitudes to treatment)
Initiation to behavioral health treatment | 6 months
  Number of participants who initiated behavioral health treatment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dartmouth College, Hanover, New Hampshire
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stecker T, Allan NP, Hoge C, Ashrafioun L, Conner KR. Efficacy of CBT for Treatment Seeking (CBT-TS) in Untreated Veterans and Service Members at Risk for Suicidal Behavior. J Gen Intern Med. 2023 Sep;38(12):2639-2646. doi: 10.1007/s11606-023-08129-z. Epub 2023 Mar 24. PMID 36964422